CLINICAL TRIAL: NCT00499421
Title: Evaluation of Intraprostatic Fiducial Markers For Targeting of External Beam Radiation Therapy
Brief Title: Evaluation of Intraprostatic Fiducial Markers For External Beam Radiation Therapy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0428
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; External Beam Radiation Therapy; Fiducial Markers; Acculoc System; Center Of Mass; EBRT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CT Scan: CT Scan with Fiducial markers + external beam radiation therapy
  Interventions: Procedure: Computed Tomography (CT) Scan

INTERVENTIONS:
Procedure: Computed Tomography (CT) Scan — CT scan of the prostate three times a week, just before the delivery of radiation.

SUMMARY:
The goal of this clinical research study is to evaluate a system for localizing (targeting for treatment) the prostate for external beam radiation therapy. The system will be used to locate the prostate before treatment and to measure movement of the prostate during treatment. The data collected with the system will be compared to CT images taken during the course of your radiation therapy treatment. Researchers will try to use this information to verify the performance of the system, which could lead to improved positioning and tracking of the prostate during treatment.

DETAILED DESCRIPTION:
The prostate may change position on a day-to-day basis due to differences in positioning, muscle tone, rectal filling, and bladder filling. Soft tissue like the prostate is not usually visible with normal x-rays, but certain metals like gold are visible. Many institutions are using an FDA-approved system (fiducial system), the one being used in this study, which involves implanting small gold markers to locate the prostate on a daily basis. This system allows the prostate to be located before treatment, which may improve radiation delivery to the prostate and decrease radiation exposure to normal tissue such as the rectum and bladder. The ability of this system to provide information on the location of the prostate before treatment should allow for more precise and accurate radiation treatment of prostate cancer.

The small implanted gold markers are 3 mm long and 1 mm wide (about the size of a grain of rice). If you agree to take part in this study, 3 markers will be permanently implanted into your prostate using a needle similar to the biopsy needle used to diagnose your cancer.

Treatment for prostate cancer during this research study will not be different from the MD Anderson standard of care. You will have intensity-modulated radiation therapy (IMRT) treatment for the prostate cancer performed using the CT-Linac treatment machine (ExaCT, Varian Medical Systems, Palo Alto, CA). This machine will have the same IMRT capabilities as other treatment machines in the Radiation Oncology Department.

During the study, the position of the gold markers seen on x-ray will be used to make adjustments to the position of your prostate for your radiation therapy treatment. The positions reported by the fiducial system will be recorded and used for daily treatment.

Three (3) times per week, you will have a CT scan of your prostate. The CT scans will be performed just before the delivery of radiation. Radiotherapists will assist you onto the treatment table and position it for your treatment. The treatment table will then be rotated 180 degrees from the treatment machine and the CT scan of your prostate will be performed. After the CT scan, which will take about 5-8 minutes, the couch will be rotated back to the original position.

A trans-abdominal ultrasound of your prostate will also be performed twice per week for the first two weeks and then once a week from then on while you are on study. The MD Anderson staff and researchers will analyze the changes in prostate movement during radiation therapy using the scanned CT images and ultrasound images and compare them with positional changes displayed by the fiducial-based system.

Targeting of your prostate on a daily basis will be performed using the fiducial-based system. This will involve performing a pair of x-rays before your treatment. A shift will be made if needed using the implanted prostate markers. The position of the seeds after the shift will be routinely verified with another pair of x-rays. After alignment has occurred, a radiation treatment will then be delivered.

This is an investigational study. The fiducial-based system is FDA-approved. A total of 20 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologic diagnosis of prostate cancer.
2. Patients must plan to have external beam radiation as the definitive treatment for their prostate cancer with daily localization.
3. Patients must be able to tolerate transrectal or transperineal implantation of three fiducial markers into the prostate.
4. Patients must be able to tolerate frequent (e.g. three CT scans per week) CT scanning.
5. Patients must be able to lie flat and still for the duration of the fiducial-based localization and CT scanning sessions.
6. Patients must have anatomy that will allow an adequate pelvic image on portal imaging and CT scanning.
7. If patients received hormone therapy, then it must have started more than 8 weeks prior to implantation of fiducials.
8. Patients on hormonal therapy at the time of simulation must remain on hormone therapy until their radiation course is complete.
9. Patients must understand and sign informed consent.

Exclusion Criteria:

1. Patients who are not candidates for trans-rectal prostate biopsy or cannot tolerate placement of three fiducial prostate markers.
2. Patients with an estimated prostate volume of less than 20 cc.
3. Patients who have had prior prostate surgery or are planned to have prostate surgery for prostate cancer.
4. Patients who have had previous radiation therapy to the pelvis.
5. Patients who have had prior prostate brachytherapy implant or who have a planned course of therapy using prostate brachytherapy (permanent seeds or high dose rate).
6. Patients with a body habitus that the CT bore of the CT/Linac treatment machine cannot accommodate (i.e. height greater than 6' 3" or body weight greater than 300 pounds).
7. Patients on anticoagulant medication (e.g., coumadin, clopidogrel, low-molecular weight heparin) other than aspirin will not be eligible. Patients on aspirin should discontinue aspirin 7 days prior to fiducial placement and for 5 days afterward.
8. Patients with hip prostheses will not be eligible.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants with prostate cancer that will be treated with external beam radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2005-09-14 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Patient Prostate Position Calculated using both fiducials and CT methods | At time of treatment planning (time 0) and at 24 additional time points during the 8-week course of radiotherapy (3 times per week)
  Prostate position determined by center of mass (COM) of prostate. COM calculated by planning system based on contours of prostate on each CT slice. Prostate position assessed as the mean position of the three implanted fiducial markers (MPIF), which is computed using software provided by the commercial fiducial system. These two points (COM and MPIF) expressed using same coordinate system, whose origin is positioned treatment isocenter. Difference between the two points (COM and MPIF) defines a vector in 3-dimensional space. The three dimensions correspond to the right-left (RL), anterior-posterior (AP), and superior-inferior (SI) directions.

CONTACTS AND LOCATIONS:
Overall Officials: Seungtaek Choi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org